CLINICAL TRIAL: NCT00178867
Title: A National Registry of Patients With Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Ravi Chari, MD, Vanderbilt University
Other Study IDs: 020116
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A registry of patients with the diagnosis of hepatocellular carcinoma.

DETAILED DESCRIPTION:
The purpose of this research is to study the factors which might cause hepatocellular carcinoma (a form of cancer arising within the liver) and compare these factors in patients from different ethnic groups and from different parts of the United States. The researchers will also conduct a survey of the stage of the cancer (how far advanced it is) and what treatments are used for this difficult-to-treat tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of hepatocellular carcinoma

Exclusion Criteria:

* Patients can not be under 18 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients seen in Hepatobiliary Surgery Clinic at Vanderbilt University Medical Center who are diagnosed with hepatocellular carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2002-01; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi S Chari, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States